CLINICAL TRIAL: NCT06273397
Title: Acetazolamide or Metolazone in Acute Heart Failure
Acronym: ACME-AHF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Alemana de Santiago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACME-AHF
Record Dates: First submitted 2024-01-31; First posted 2024-02-22 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure Acute; Decompensated Heart Failure
Keywords: Acetazolamide; Metolazone; Heart Failure Acute
MeSH Terms: interventions — Acetazolamide; Metolazone; Furosemide

STUDY DESIGN:
Intervention Model Description: This is an Open, Multicenter, Prospective, and Randomized study with three treatment arms. The outcomes to be assessed in the initial phase will be at 4 days post-randomization, followed by evaluation at 90 days after hospital discharge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Furosemide alone (Active Comparator): Active comparator arm with intravenous furosemide dosing based on glomerular filtration rate (protocol).
  Interventions: Drug: Furosemide Injection
- Acetazolamide plus Furosemide (Experimental): Experimental arm number 1 corresponds to oral acetazolamide 250mg (once daily) in combination with furosemide according to the protocol.
  Interventions: Drug: Acetazolamide 250 MG; Drug: Furosemide Injection
- Metolazone plus Furosemide (Experimental): Experimental arm number 2 corresponds to oral metolazone 2.5mg (once daily) in combination with furosemide according to the protocol.
  Interventions: Drug: Metolazone 2.5 MG; Drug: Furosemide Injection

INTERVENTIONS:
Drug: Acetazolamide 250 MG — Acetazolamide 250mg orally per day plus furosemide as per protocol. The intervention is administered on the day of hospital admission and for two consecutive mornings. The total intervention consists of 3 doses. The intervention is discontinued on the third morning. The calculation of the congestion score is performed every morning until the third morning. If complete decongestion is achieved, the primary outcome will be considered fulfilled.
  Arms: Acetazolamide plus Furosemide
Drug: Metolazone 2.5 MG — Metolazone 2.5mg orally per day plus furosemide as per protocol. The intervention is administered on the day of hospital admission and for two consecutive mornings. The total intervention consists of 3 doses. The intervention is discontinued on the third morning. The calculation of the congestion score is performed every morning until the third morning. If complete decongestion is achieved, the primary outcome will be considered fulfilled.
  Arms: Metolazone plus Furosemide
Drug: Furosemide Injection — Intravenous furosemide in a double daily dose. The dosage is determined by a predefined table based on the admission renal function and the outpatient dose prior to admission. In general terms, for patients with an estimated glomerular filtration rate above 60 ml/min/1.73m² or those experiencing heart failure debut, the dose will be 1x the outpatient dose. For those with a glomerular filtration rate below 60 ml/min/1.73m², the dose will be 2x the outpatient dose. The dosing protocol for this arm also serves as guidance for furosemide in the intervention arms.

SUMMARY:
Impact of Acute Heart Failure:

According to the World Health Organization (WHO), approximately 26 million people suffer from Heart Failure (HF), with a mortality rate of up to 50% within five years of diagnosis. Acute Heart Failure (AHF) exacerbations, leading to hospitalization, are common and represent the primary cause of hospital admissions in those over 65. Effective decongestion during hospitalization is crucial, as failure to achieve it doubles the risk of rehospitalization and mortality, incurring significant healthcare costs.

Use of Diuretics in Acute Heart Failure:

Diuretics, particularly loop diuretics like furosemide, are a cornerstone in managing AHF by inducing natriuresis and achieving decongestion. Clinical experience supports their use, though limited clinical trials exist. Pharmacological concepts guide their administration, emphasizing intravenous delivery in high doses and adjusting subsequent doses based on decongestive efficacy. Additionally, sequential tubular blockade with other diuretics like metolazone and acetazolamide is explored to enhance decongestion.

Use of Metolazone and Acetazolamide:

Sequential tubular blockade, using metolazone and acetazolamide in conjunction with furosemide, aims to achieve rapid and effective decongestion. While metolazone targets the distal tubule, inhibiting sodium-chloride channels, acetazolamide affects proximal tubular function. Studies like ADVOR (acetazolamide) and CLOROTIC (thiazide-like diuretic) demonstrate the potential benefits of combining these diuretics for quicker decongestion but with potential risks (in the case of Hydrochlorothiazide).

Outcomes Measured by Major Studies:

Recent studies assessing decongestion in AHF reveal a lack of uniformity in outcome selection. The primary focus should be on reducing rehospitalizations and post-discharge mortality by achieving effective decongestion. The ADVOR study, using a simple congestion score based on clinical and imaging criteria, underscores the importance of reaching a congestion score of 0 or 1 promptly.

Congestion Monitoring:

Monitoring diuretic treatment solely based on clinical aspects may not capture subclinical congestion, necessitating biochemical and imaging parameters. The ACME-AHF trial proposes a diagnostic score integrating clinical and imaging aspects to evaluate congestion status. Secondary outcomes include cumulative diuresis, weight loss, diuretic efficiency, and natriuresis, with a focus on natriuresis as a reliable physiological parameter for decongestion.

Aim of the study:

The ACME-AHF trial is designed to compare the efficacy and safety of two diuretic combination strategies: acetazolamide with furosemide and metolazone with furosemide. The primary objective is to relieve congestion, assessed using a congestion score, within the first three days of treatment during an hospitalization for acute heart failure.

DETAILED DESCRIPTION:
After inclusion in the study and signing the informed consent, the patient will be randomized into one of the following three intervention groups:

* Group A: Intravenous furosemide alone.
* Group B: Intravenous furosemide with oral metolazone 2.5mg.
* Group C: Intravenous furosemide with oral acetazolamide 250mg.

Metolazone or acetazolamide will be administered in fixed doses for a total of 3 doses (D0, D1, and D2) - at admission (D0), on the morning of the second day (D1), and on the morning of the third day (D2).

The use of intravenous furosemide will follow a protocol for dose and frequency of administration. Its dose should not be modified before D2. On D2, modification is allowed according to the protocol (details later).

In cases of major adverse events only, the local practitioner may suspend these therapies (as indicated later).

The study is driven by a clinical outcome based on a congestion score. The primary outcome will assess the ability to achieve effective decongestion (score 0 - 1) for each of the three interventions over 3 days. The primary outcome will be considered achieved if a score of 0 - 1 is reached on D1, D2, or D3, without requiring escalation of diuretic therapy on D2. The congestion score consists of 3 clinical parameters (edema, jugular venous distension, lung crepitations), one radiological parameter (pleural effusion on X-ray), and one ultrasonographic parameter (LUS: B-line count in 4 zones). A score is assigned based on the intensity of each parameter, with 0 and 1 considered as a score indicative of complete decongestion.

The key determinant on D0, D1, and D2, guiding whether the intervention continues or stops, is the persistence of congestion. The intervention should continue for those with a congestion score of 2 or more during the first assessment of the day. If the congestion score is 0 or 1, the intervention is suspended, and the patient should transition to oral furosemide (in preparation for hospital discharge).

Here is the detailed procedure for each day of intervention (total 3 days, closing on the third morning of hospitalization or D3):

* D0 or admission day: Eligibility criteria are reviewed for study inclusion, informed consent is obtained, and randomization to the intervention arm is conducted. Admission data is collected.
* D1 or first morning after admission: Congestion score is calculated. In case the primary outcome is not achieved, the intervention continues without modifications. Clinical and biochemical data are collected according to the protocol.
* D2 or second morning of hospitalization: Congestion score is calculated, and the intervention continues in case the primary outcome is not achieved. On this day, decongestive therapy is titrated based on the total diuresis and weight loss achieved in the previous 24 hours (according to the protocol).
* D3 or third morning: Congestion score is calculated. The intervention is discontinued regardless of the achieved score. Further management is at the discretion of the treating physician. Clinical and biochemical data for the last day are collected.
* 90-day Follow-up: The patient will be contacted, and the medical records will be reviewed to assess clinical and biochemical data 90 days after discharge. Information on worsening heart failure and mortality during this period will be extracted.

Additional recommendations for the intervention include:

1. Optimal Medical Treatment: Maintain chronic heart failure therapy (ACEI/ARNI/ARB, Beta-blockers, Mineralocorticoid receptor antagonists, and SGLT2 inhibitors) unless contraindicated. Initiate these treatments before discharge, if not already instituted. Encourage early medical follow-up for discharged patients. Decisions on ferric carboxymaltose administration and entry into cardiac rehabilitation are at the physician's discretion.
2. Potassium Control: Suggested to keep plasma levels above 4.0 mEQ/L (oral or intravenous correction).
3. Patient Diet and Mobilization: Recommend restricting sodium and volume to less than 1.5g and 2000cc daily, respectively. Encourage early mobilization and kinesiotherapy, if no contraindications. Provide thromboembolic prevention based on local guidelines.
4. Situations for Intervention Cessation: (protocol termination and AE reporting)

   * Hypokalemia < 2.5 mEQ/L
   * Hyponatremia < 125 mEQ/L
   * Acidosis with pH < 7.20 or Bicarbonate < 15 mEQ/L
   * Asymptomatic hypotension (SBP < 90mmHg) or symptomatic hypotension (SBP < 100mmHg).
   * Significant deterioration in renal function (creatinine rise above 0.8mg and 1.5x baseline) NOTE: If early intervention suspension occurs with complete decongestion, consider the primary outcome achieved.

ELIGIBILITY:
Inclusion Criteria:

* Acute heart failure: Hospitalization due to symptoms of heart failure, congestion signs documented with a congestion score greater than 1, NT-proBNP above 1000 pg/ml.
* Randomization within 24 hours of admission.

Exclusion Criteria:

* Under 18 years of age.
* Received more than one dose of intravenous furosemide before randomization.
* Cause of heart failure: hypertrophic or restrictive cardiomyopathy, or constrictive pericarditis.
* Acute coronary syndrome or severe acute valvulopathy as the cause of decompensation.
* Systolic blood pressure < 90mmHg before randomization.
* Requirement for vasopressors, inotropes, or invasive mechanical ventilation. Use of intravenous vasodilators or non-invasive mechanical ventilation is allowed.
* Glomerular filtration rate < 20ml/min/1.73m2.
* Potassium < 2.5 mEQ/L or Sodium < 125 mEQ/L before randomization.
* pH < 7.2 or Bicarbonate < 15mEQ/L before randomization.
* Use of another diuretic in addition to furosemide before randomization. Dapagliflozin or Empagliflozin can be maintained upon admission or initiated early during hospitalization if desired by the treating physician (variable to be recorded).
* Patients who cannot achieve adequate recording of variables (e.g., inability to quantify diuresis or weight).
* Pregnant or lactating individuals. If of childbearing age and there is inconsistency with contraceptive use or reasonable doubts about current pregnancy, a pregnancy test must be conducted before study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Treatment success | 4 days
  Complete decongestion by the third morning without requiring escalation in diuretic therapy (by the second morning).

SECONDARY OUTCOMES:
Mortality | 3 months
  All-cause mortality during the first 3 months after start of the study
Worsening Heart Failure | 3 months
  Readmission for Heart Failure or Urgent visit for Heart Failure during the first 3 months after start of the study
Cumulative 24-hour Natriuresis | Day 2
  Natriuresis measured on the second day
Cumulative weight loss | 4 days
  Cumulative weight loss by the third morning
Subclinical congestion | 4 days
  Congestion score will be the score used in the study to evaluate the primary outcome. The calculated scores can range from 0 to 12 points, with 0 indicating absence of congestion and 12 representing the highest degree of congestion. The primary outcome will be defined as achieving a score of 0 or 1 and also having absence of B-lines in the lung ultrasound (negative LUS criterion). In this secondary outcome, the presence of subclinical congestion will be evaluated, which is defined as a congestion score of 0 or 1 but with a positive LUS.
Change in Hematocrit value | 4 days
  Change in Hematocrit
Change in NT-proBNP concentration | 4 days
  Change in NT-proBNP
Change in CA125 value | 4 days
  Change in CA125

OTHER OUTCOMES:
Any adverse event | 3 months
  Any adverse clinical event related to intervention during the first 3 months after start of the study
Changes in pH value | 4 days
  Change in pH over the specified time period
Change in plasma electrolyte values | 4 days
  Change in plasma concentration of sodium, potassium, and chloride

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rivas-Lasarte M, Maestro A, Fernandez-Martinez J, Lopez-Lopez L, Sole-Gonzalez E, Vives-Borras M, Montero S, Mesado N, Pirla MJ, Mirabet S, Fluvia P, Brossa V, Sionis A, Roig E, Cinca J, Alvarez-Garcia J. Prevalence and prognostic impact of subclinical pulmonary congestion at discharge in patients with acute heart failure. ESC Heart Fail. 2020 Oct;7(5):2621-2628. doi: 10.1002/ehf2.12842. Epub 2020 Jul 7. PMID 32633473
- [Background] Urbich M, Globe G, Pantiri K, Heisen M, Bennison C, Wirtz HS, Di Tanna GL. A Systematic Review of Medical Costs Associated with Heart Failure in the USA (2014-2020). Pharmacoeconomics. 2020 Nov;38(11):1219-1236. doi: 10.1007/s40273-020-00952-0. PMID 32812149
- [Background] Felker GM, Ellison DH, Mullens W, Cox ZL, Testani JM. Diuretic Therapy for Patients With Heart Failure: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Mar 17;75(10):1178-1195. doi: 10.1016/j.jacc.2019.12.059. PMID 32164892
- [Background] Felker GM, Lee KL, Bull DA, Redfield MM, Stevenson LW, Goldsmith SR, LeWinter MM, Deswal A, Rouleau JL, Ofili EO, Anstrom KJ, Hernandez AF, McNulty SE, Velazquez EJ, Kfoury AG, Chen HH, Givertz MM, Semigran MJ, Bart BA, Mascette AM, Braunwald E, O'Connor CM; NHLBI Heart Failure Clinical Research Network. Diuretic strategies in patients with acute decompensated heart failure. N Engl J Med. 2011 Mar 3;364(9):797-805. doi: 10.1056/NEJMoa1005419. PMID 21366472
- [Background] Mullens W, Dauw J, Martens P, Verbrugge FH, Nijst P, Meekers E, Tartaglia K, Chenot F, Moubayed S, Dierckx R, Blouard P, Troisfontaines P, Derthoo D, Smolders W, Bruckers L, Droogne W, Ter Maaten JM, Damman K, Lassus J, Mebazaa A, Filippatos G, Ruschitzka F, Dupont M; ADVOR Study Group. Acetazolamide in Acute Decompensated Heart Failure with Volume Overload. N Engl J Med. 2022 Sep 29;387(13):1185-1195. doi: 10.1056/NEJMoa2203094. Epub 2022 Aug 27. PMID 36027559
- [Background] Trullas JC, Morales-Rull JL, Casado J, Carrera-Izquierdo M, Sanchez-Marteles M, Conde-Martel A, Davila-Ramos MF, Llacer P, Salamanca-Bautista P, Perez-Silvestre J, Plasin MA, Cerqueiro JM, Gil P, Formiga F, Manzano L; CLOROTIC trial investigators. Combining loop with thiazide diuretics for decompensated heart failure: the CLOROTIC trial. Eur Heart J. 2023 Feb 1;44(5):411-421. doi: 10.1093/eurheartj/ehac689. PMID 36423214
- [Background] Appiani F. [Monitoring decongestion in acute heart failure]. Rev Med Chil. 2022 Apr;150(4):493-504. doi: 10.4067/S0034-98872022000400493. Spanish. PMID 36155759